CLINICAL TRIAL: NCT01470378
Title: Manual Lymphatic Drainage in Women Undergone to Thigh Lifting After Bariatric Surgery
Brief Title: Manual Lymphatic Drainage in Women Undergone to Thigh Lifting
Acronym: Thight_lift
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Lilia Cristina de Arruda, Principal Investigator, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UNIFESP_LILIA
Record Dates: First submitted 2011-11-02; First posted 2011-11-11 (Estimated); Last update posted 2013-08-09 (Estimated); Status verified 2013-08

CONDITIONS: Lymphedema; Obesity
Keywords: Lymphedema; Magnetic Resonance Imaging; Plastic Surgery
MeSH Terms: conditions — Lymphedema; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Group (Active Comparator): This group will not be undergoing to manual lymphatic drainage
  Interventions: Procedure: Thigh Surgery
- Study Group (Active Comparator): This group will be undergoing to manual lymphatic drainage
  Interventions: Procedure: Thigh Surgery

INTERVENTIONS:
Procedure: Thigh Surgery — Circumferential thigh surgery post bariatric surgery
  Other Names: Thigh plastic surgery; Postobesity surgery

SUMMARY:
This study will investigate the subcutaneous tissue changes in the lymphedema found after thigh surgery, by circumferential measure of thr thighs and by magnetic resonance imaging verifying the effects of postoperative lymphatic drainage.

DETAILED DESCRIPTION:
Patients will be invited to participate in the study, divided into two groups, and randomized to treatment by wwww.randomization.com, where 10 patients will participate in the study group(20 legs) and 10 control group patients(20 legs). Total of 40 legs. Then, the evaluation will be performed on preoperative time, consisting of physical examination and circumferential measures. Others measurements will be taken im postoperative time and confirmed by magnetic resonance.

ELIGIBILITY:
Inclusion Criteria:

* Female patients
* Age between 30 and 60 years old
* Bariatric Surgery Capella Previous Type
* Stabilization of weight loss for 1 year or more
* Patients with a body mass index less than or equal to 30 kg/m2

Exclusion Criteria:

* Pregnancy, childbirth or breastfeeding for less than 1 year
* Presence of uncontrolled systemic disease
* Other disease that require surgical interventions
* Lymphatic or venous pathologies in advance
* Patients over 110 kg
* Patients with a body mass index(BMI) greater than 30 kg/m2
* Patients who has undergone plastic surgery of the thighs

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-11 (Actual); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
Preoperative measurement. | one day before surgery
  Thigh circumference measurements made with anthropometric metal tape and a Permanent Marker, based in bone parameters in supine position. Using as reference the bony protuberance of the trochanter, the first measurement will be taken 5 (five) cm below this point and 5 (five) cm above the patella, and betwin this two points will be made one mark at the midpoint between them. After the measurement, a Magnetic Resonance of the thighs is made.

SECONDARY OUTCOMES:
Thighs circumference measurement | 7th postoperative day
  Thigh circumference measurements made with anthropometric metal tape and a Permanent Marker, based in bone parameters in supine position. Using as reference the bony protuberance of the trochanter, the first mesurement will be taken 5 (five) cm below this point and 5 (five) cm above the patella, and betwin this two points will be made one mark at the midpoint between them
Thighs circumference measurement | 9th postoperative day
  Thigh circumference measurements made with anthropometric metal tape and a Permanent Marker, based in bone parameters in supine position. Using as reference the bony protuberance of the trochanter, the first mesurement will be taken 5 (five) cm below this point and 5 (five) cm above the patella, and betwin this two points will be made one mark at the midpoint between them
Thighs circumference measurement | 14th postoperative day
  Thigh circumference measurements made with anthropometric metal tape and a Permanent Marker, based in bone parameters in supine position. Using as reference the bony protuberance of the trochanter, the first mesurement will be taken 5 (five) cm below this point and 5 (five) cm above the patella, and betwin this two points will be made one mark at the midpoint between them. After the measurement, a Magnetic Resonance of the thighs is made.
Thighs circumference measurement | 16th postoperative day
  Thigh circumference measurements made with anthropometric metal tape and a Permanent Marker, based in bone parameters in supine position. Using as reference the bony protuberance of the trochanter, the first mesurement will be taken 5 (five) cm below this point and 5 (five) cm above the patella, and betwin this two points will be made one mark at the midpoint between them.
Thighs circumference measurement | 21th postoperative day
  Thigh circumference measurements made with anthropometric metal tape and a Permanent Marker, based in bone parameters in supine position. Using as reference the bony protuberance of the trochanter, the first mesurement will be taken 5 (five) cm below this point and 5 (five) cm above the patella, and betwin this two points will be made one mark at the midpoint between them.
Thighs circumference measurement | 28th postoperative day
  Thigh circumference measurements made with anthropometric metal tape and a Permanent Marker, based in bone parameters in supine position. Using as reference the bony protuberance of the trochanter, the first mesurement will be taken 5 (five) cm below this point and 5 (five) cm above the patella, and betwin this two points will be made one mark at the midpoint between them. After the measurement, a Magnetic Resonance of the thighs is made.

CONTACTS AND LOCATIONS:
Overall Officials: Lydia M Ferreira, MD, Study Chair — Federal University of São Paulo
Locations (1):
- Federal University of Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Le Louarn C, Pascal JF. The concentric medial thigh lift. Aesthetic Plast Surg. 2004 Jan-Feb;28(1):20-3. doi: 10.1007/s00266-003-3095-x. Epub 2004 Mar 25. PMID 15037958
- [Background] Nemerofsky RB, Oliak DA, Capella JF. Body lift: an account of 200 consecutive cases in the massive weight loss patient. Plast Reconstr Surg. 2006 Feb;117(2):414-30. doi: 10.1097/01.prs.0000197524.18233.bb. PMID 16462321
- [Background] Pascal JF, Le Louarn C. Remodeling bodylift with high lateral tension. Aesthetic Plast Surg. 2002 May-Jun;26(3):223-30. doi: 10.1007/s00266-002-1478-z. PMID 12140705
- [Background] Moreno CH, Neto HJ, Junior AH, Malheiros CA. Thighplasty after bariatric surgery: evaluation of lymphatic drainage in lower extremities. Obes Surg. 2008 Sep;18(9):1160-4. doi: 10.1007/s11695-007-9400-z. Epub 2008 Jun 11. PMID 18546051
- [Background] Kolker AR, Xipoleas GD. The circumferential thigh lift and vertical extension circumferential thigh lift: maximizing aesthetics and safety in lower extremity contouring. Ann Plast Surg. 2011 May;66(5):452-6. doi: 10.1097/SAP.0b013e3182145682. PMID 21451373
- See also: The Obesity Society is the leading scientific society dedicated to the study of obesity — http://www.obesity.org/
- See also: OBESITY - ONLINE is a multi-disciplinary forum for research and treatment of massive obesity, including plastics, psychiatry, endocrinology, nutrition, nursing, dietetics and allied health — http://www.obesity-online.com/